CLINICAL TRIAL: NCT00856310
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study of the Safety and Tolerability of REGN475 in Healthy Subjects
Brief Title: A Single-Dose Study of the Safety and Tolerability of REGN475(SAR164877) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R475-PN-0817
Record Dates: First submitted 2009-02-12; First posted 2009-03-05 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Active Comparator): Dose 1 REGN475
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 2 (Active Comparator): Dose 2 of REGN475
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 3 (Active Comparator): Dose 2 of REGN475
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 4 (Active Comparator): Dose 1 of REGN475
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 5 (Active Comparator): Dose 2 of REGN475
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 6 (Active Comparator): Dose 1 REGN475 subcutaneous administration
  Interventions: Biological: REGN475 (SAR164877)
- Cohort 7 (Active Comparator): Dose 2 REGN475 subcutaneous administration
  Interventions: Biological: REGN475 (SAR164877)

INTERVENTIONS:
Biological: REGN475 (SAR164877) — Subcutaneous administration REGN475 (SAR164877)

SUMMARY:
This is a randomized, double-blind, placebo-controlled single-dose study of the safety and tolerability of intravenously administered REGN475 in healthy volunteers. The primary objective of the study is to assess the safety and tolerability of REGN475. The secondary objectives are to characterize the pharmacokinetic and immunogenicity profiles of REGN475.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female volunteers, in general good health and 21 to 65 years of age.
* Female volunteers must be post-menopausal for at least 1 year or surgically sterile.

Key Exclusion Criteria:

* Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, GI, hepatic, metabolic or lymphatic disease that would adversely affect the subject's participation in this study or interpretation of safety/ PK data
* Participation in any clinical research study evaluating another investigational drug or therapy within 3 weeks or at least 5 half-lives of the investigational drug, whichever is longer, prior to the Screening Visit.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events in subjects treated with REGN475 or placebo. | 16 weeks

SECONDARY OUTCOMES:
Serum concentrations of REGN475. | 16 Weeks
The presence or absence of antibodies against REGN475. | 16 Week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Altoona, Pennsylvania, United States